CLINICAL TRIAL: NCT01397422
Title: Extended Release Amantadine Safety and Efficacy Study in Levodopa-Induced Dyskinesia (EASED Study)
Acronym: EASED
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Adamas Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADS-PAR-AM201
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Dyskinesia; Levodopa Induced Dyskinesia; Parkinson's Disease
Keywords: Levodopa-induced dyskinesia; Parkinsonism
MeSH Terms: conditions — Dyskinesias; Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment A (Placebo Comparator)
  Interventions: Drug: ADS-5102 (extended release amantadine HCl)
- Treatment B (Active Comparator): Low dose ADS-5102 (amantadine extended release)
  Interventions: Drug: ADS-5102 (extended release amantadine HCl)
- Treatment C (Active Comparator): A mid-dose ADS-5102 (amantadine extended release)
  Interventions: Drug: ADS-5102 (extended release amantadine HCl)
- Treatment D (Active Comparator): High dose ADS-5102 (amantadine extended release)
  Interventions: Drug: ADS-5102 (extended release amantadine HCl)

INTERVENTIONS:
Drug: ADS-5102 (extended release amantadine HCl) — Oral capsules to be administered once daily at bedtime, for 8 weeks

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, 4-arm parallel group study to evaluate the tolerability and efficacy of each of three dose levels of ADS-5102 oral capsules, an extended release formulation of amantadine, dosed once daily for the treatment of levodopa-induced dyskinesia (LID) in subjects with Parkinson's disease (PD). The novel pharmacokinetic profile of ADS-5102 is expected to achieve i) higher amantadine plasma concentrations during daytime hours when dyskinesia as well as motor and non-motor symptoms of PD are most problematic, ii) low amantadine plasma concentrations overnight, which may reduce the sleep disturbances and vivid dreams occasionally associated with amantadine, and iii) a reduced initial rate of rise in plasma concentration, which is expected to improve overall tolerability of amantadine.

ELIGIBILITY:
Inclusion Criteria:

* Signed a current IRB/IEC-approved informed consent form
* Parkinson's disease, per UK Parkinson's Disease Society (UKPDS) Brain Bank Clinical Diagnostic Criteria
* On a stable regimen of antiparkinson's medications , including any levodopa preparation administered not less than three times daily, and willing to continue the same doses and regimens during study participation
* Experiencing troublesome dyskinesia following levodopa dosing (peak dose dyskinesia)
* Able to understand and complete a standardized PD home diary, following training

Exclusion Criteria:

* History of neurosurgical intervention related to Parkinson's disease (e.g. deep brain stimulation)
* History of seizures or stroke/TIA within 2 years of screening
* History of cancer within 5 years of screening, except adequately treated non-melanomatous skin cancers, localized bladder cancer, non-metastatic prostate cancer or in situ cervical cancer
* Estimated GFR < 50 mL/min/1.73m2
* Presence of cognitive impairment, as evidenced by a Mini-Mental Status Examination (MMSE) score of less than 24 during screening
* If female, is pregnant or lactating, or has a positive pregnancy test result pre-dose
* If a sexually active female, is not surgically sterile or at least 2 years post-menopausal, or does not agree to utilize an effective method of contraception from screening through at least 4 weeks after the completion of study treatment
* Treatment with an investigational drug or device within 30 days prior to screening
* Treatment with an investigational biologic within 6 months prior to screening

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Director, Study Director — Adamas Pharmaceuticals, Inc.
Locations (33):
- United States (33):
  - Sun City, Arizona
  - Fountain Valley, California
  - Long Beach, California
  - Los Angeles, California
  - Oxnard, California
  - Pasadena, California
  - Reseda, California
  - Sunnyvale, California
  - Ventura, California
  - Fairfield, Connecticut
  - Boca Raton, Florida
  - Bradenton, Florida
  - Port Charlotte, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Winfield, Illinois
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Boston, Massachusetts
  - West Bloomfield, Michigan
  - Toms River, New Jersey
  - New York, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Houston, Texas
  - San Antonio, Texas
  - Richmond, Virginia
  - Kirkland, Washington
  - Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Parkinson's disease (PD) and Levodopa-induced Dyskinesia (LID) were enrolled at 31 study sites in the United States. The first subject was randomized on 03 August 2011 and the last subject completed on 15 April 2013.
Pre-assignment Details: All randomized subjects (83) were treated and analyzed for safety; 80 were analyzed for efficacy and included in the Modified Intent to Treat (MITT) population. Subjects in the MITT had mild to severe dyskinesia, had periods of troublesome dyskinesia during the day, received ≥ 1 dose of study drug, and provided ≥ 1 postbaseline efficacy assessment.
Groups:
- Placebo: ADS-5102 matching placebo: oral capsules administered once daily at bedtime for 8 weeks
- ADS-5102 (260 mg): 260 mg dose of ADS-5102 (amantadine HCl extended release): oral capsules administered once daily at bedtime for 8 weeks
- ADS-5102 (340 mg): 340 mg dose of ADS-5102 (amantadine HCl extended release): oral capsules administered once daily at bedtime for 8 weeks (260 mg Week 1; 340 mg Weeks 2-8)
- ADS-5102 (420 mg): 420 mg dose of ADS-5102 (amantadine HCl extended release): oral capsules administered once daily at bedtime for 8 weeks (260 mg Week 1; 340 mg Week 2; 420 mg Weeks 3-8)
Period: Overall Study
Arm/Group | Placebo | ADS-5102 (260 mg) | ADS-5102 (340 mg) | ADS-5102 (420 mg)
Started | 22 | 20 | 21 (Of the 3 participants who discontinued, 1 withdrew due to both an AE and an eGFR < 50 mL/min/1.73m^2) | 20
Completed | 20 | 17 | 18 (AE = adverse event; eGFR = estimated glomerular filtration rate) | 12
Not Completed | 2 | 3 | 3 | 8
Not completed — Adverse Event | 0 | 3 | 3 | 8
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Increased bradykinesia related to PD | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population (all randomized subjects who received ≥ 1 dose of study drug)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ADS-5102 (260 mg) | ADS-5102 (340 mg) | ADS-5102 (420 mg) | Total
Number analyzed (Participants) | 22 | 20 | 21 | 20 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (10.17) | 67.5 (8.59) | 64.7 (10.03) | 66.4 (9.38) | 66.0 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 8 | 10 | 38
  Male | 14 | 8 | 13 | 10 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 2 | 5
  Not Hispanic or Latino | 21 | 18 | 21 | 18 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 2
  Asian | 1 | 0 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 20 | 18 | 20 | 17 | 75
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Fatigue Severity Score (FSS) [Mean (Standard Deviation); unit: units on a scale] — The FSS is a 9-item self-reported scale, rating subject experience of fatigue during the previous 7 days. The total score, on a scale from 1-7, is represented by the mean of all answered items. The higher the score, the greater the fatigue severity.
  units on a scale | 4.86 (1.211) | 4.40 (1.488) | 4.80 (1.425) | 4.78 (1.120) | 4.71 (1.307)
Hoehn and Yahr Score [Mean (Standard Deviation); unit: units on a scale] — Hoehn and Yahr assessed at screening only. The scale, from 1-5, describes the patient's PD progression. The higher the score the more severe the symptoms of PD.
  units on a scale | 2.5 (0.7) | 2.5 (0.9) | 2.5 (0.6) | 2.4 (0.8) | 2.5 (0.7)
Time since PD diagnosis [Mean (Standard Deviation); unit: years] | 10.66 (7.057) | 8.94 (3.395) | 9.33 (4.913) | 9.00 (3.484) | 9.51 (4.964)
Levodopa daily dose [Mean (Standard Deviation); unit: mg] | 801.1 (431.94) | 714.5 (449.33) | 694.0 (278.33) | 862.5 (585.94) | 768.6 (444.41)
Duration of LID [Mean (Standard Deviation); unit: years] | 4.08 (4.051) | 3.35 (2.585) | 4.37 (3.364) | 3.57 (2.049) | 3.85 (3.106)
Subjects taking Antiparkinson Medication [Count of Participants; unit: Participants] — Participants may have been taking more than 1 antiparkinson medication at baseline.
  Participants
    Levodopa (Sinemet or Stalevo) | 22 | 20 | 21 | 20 | 83
    Dopamine Agonist | 14 | 14 | 10 | 16 | 54
    MAO-B Inhibitor | 14 | 11 | 12 | 12 | 49
    COMT Inhibitor | 3 | 1 | 6 | 4 | 14
    Anticholinergic | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in the Unified Dyskinesia Rating Scale (UDysRS) Total Score From Baseline to Week 8
Description: The UDysRS is a dyskinesia rating scale from 0-104, and it evaluates involuntary movements associated with PD. A higher score indicates more severe PD. The last observation carried forward (LOCF) method was used for analysis. Participants were summarized according to the actual treatment received.
Time Frame: Baseline (Day 1) and Week 8
Population: Participants in the MITT population with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- ADS-5102 (260 mg): 260 mg dose of ADS-5102 (amantadine HClextended release): oral capsules administered once daily at bedtime for 8 weeks
- ADS-5102 (420 mg): 420 mg dose of ADS-5102 (amantadine HClextended release): oral capsules administered once daily at bedtime for 8 weeks (260 mg Week 1; 340 mg Week 2; 420 mg Weeks 3-8)
Arm/Group | Placebo | ADS-5102 (260 mg) | ADS-5102 (340 mg) | ADS-5102 (420 mg)
Number analyzed (Participants) | 22 | 19 | 20 | 19
units on a scale | -6.7 (2.68) | -12.3 (2.88) | -17.9 (2.82) | -16.7 (2.88)
Statistical Analysis 1: Comparison: ADS-5102 (340 mg); 20 subjects per treatment arm provided 80% power using a 2-sided 2-sample test at 5% significance. The null hypothesis for the primary endpoint was that the response of the ADS-5102 340 mg group was equal to that of the placebo group; Test type: Superiority; p = 0.0051, ANCOVA; Change from baseline is a dependent variable, treatment group is a factor, and the baseline value is a covariate; Least Squares Mean Difference = -11.3, 95% CI 2-sided [-19.1 to -3.5]
Statistical Analysis 2: Comparison: ADS-5102 (420 mg); Test type: Superiority; p = 0.0131, ANCOVA; Least Squares Mean Difference = -10.0, 95% CI 2-sided [-17.8 to -2.2]
Statistical Analysis 3: Comparison: ADS-5102 (260 mg); Test type: Superiority; p = 0.1595, ANCOVA; Least Squares Mean Difference = -5.6, 95% CI 2-sided [-13.4 to 2.2]

2. Secondary Outcome: Change in the Fatigue Severity Score (FSS) From Baseline to Week 8
Description: The FSS is a 9-item self-reported scale, rating subject experience of fatigue during the previous 7 days. The total score, on a scale from 1-7, is represented by the mean of all answered items. The higher the score, the greater the fatigue severity.
Time Frame: Baseline (Day 1) and Week 8
Population: MITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ADS-5102 (260 mg) | ADS-5102 (340 mg) | ADS-5102 (420 mg)
Number analyzed (Participants) | 22 | 19 | 20 | 19
units on a scale | -0.25 (0.267) | -0.06 (0.289) | -0.55 (0.280) | 0.00 (0.287)
Statistical Analysis 1: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.4314, ANCOVA; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-1.1 to 0.5]
Statistical Analysis 2: Comparison: ADS-5102 (420 mg); Test type: Superiority; p = 0.5223, ANCOVA; Least Squares Mean Difference = 0.3, 95% CI 2-sided [-0.5 to 1.0]
Statistical Analysis 3: Comparison: ADS-5102 (260 mg); Test type: Superiority; p = 0.6298, ANCOVA; Change from baseline is a dependent variable, treatment group is a factor, baseline value is a covariate; Least Squares Mean Difference = 0.2, 95% CI 2-sided [-0.6 to 1.0]

3. Secondary Outcome: Change in Total Objective Score (III, IV) of the UDysRS From Baseline to Week 8
Description: UDysRS Part III measures objective impairment (dyskinesia severity, anatomic distribution, and type, based on 4 observed activities); and Part IV measures objective disability based on Part III activities. The scores for the 2 Parts combined range from 0-44; a higher score represents more severe dyskinesia.
Time Frame: Baseline (Day 1) and Week 8
Population: MITT Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ADS-5102 (260 mg) | ADS-5102 (340 mg) | ADS-5102 (420 mg)
Number analyzed (Participants) | 22 | 19 | 20 | 19
units on a scale | -1.9 (1.19) | -4.4 (1.26) | -7.1 (1.24) | -8.3 (1.26)
Statistical Analysis 1: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.0038, ANCOVA; Least Squares Mean Difference = -5.2, 95% CI 2-sided [-8.7 to -1.7]
Statistical Analysis 2: Comparison: ADS-5102 (420 mg); Test type: Superiority; p = 0.0004, ANCOVA; Least Squares Mean Difference = -6.4, 95% CI 2-sided [-9.8 to -2.9]
Statistical Analysis 3: Comparison: ADS-5102 (260 mg); Test type: Superiority; p = 0.1469, ANCOVA; Change from baseline is a dependent variable, treatment group is a factor, and the baseline value is a covariate; Least Squares Mean Difference = -2.5, 95% CI 2-sided [-6.0 to 0.9]

4. Secondary Outcome: Change in ON Time Without Troublesome Dyskinesia (ON Without Dyskinesia Plus ON With Non-troublesome Dyskinesia) From Baseline to Week 8; Based on a Standardized PD Home Diary
Description: A PD home diary was used to score 5 different conditions in 30-minute time intervals: ASLEEP, OFF, ON (ie, had adequate control of PD symptoms) without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia. The results were based on 2 consecutive 24-hour diaries taken prior to the day of randomization and prior to the Week 8 visit.
Time Frame: Baseline (Day 1) and Week 8
Population: MITT population
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | ADS-5102 (260 mg) | ADS-5102 (340 mg) | ADS-5102 (420 mg)
Number analyzed (Participants) | 22 | 19 | 20 | 19
hours | 0.9 (0.76) | 4.1 (0.82) | 3.8 (0.79) | 3.6 (0.83)
Statistical Analysis 1: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.0078, ANCOVA; Least Squares Mean Difference = 3.0, 95% CI 2-sided [0.8 to 5.2]
Statistical Analysis 2: Comparison: ADS-5102 (420 mg); Test type: Superiority; p = 0.0179, ANCOVA; Least Squares Mean Difference = 2.7, 95% CI 2-sided [0.5 to 5.0]
Statistical Analysis 3: Comparison: ADS-5102 (260 mg); Test type: Superiority; p = 0.0040, ANCOVA; Change from baseline is a dependent variable, treatment group is a factor, and the baseline value is a covariate; Least Squares Mean Difference = 3.3, 95% CI 2-sided [1.1 to 5.5]

5. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Combined Scores (Parts I, II, III) From Baseline to Week 8
Description: The MDS-UPDRS Parts I, II, and III examined non-motor experiences of daily living, motor experiences of daily living, and motor examination, respectively. Each part had sub scales ranging from normal = 0 to severe = 4.
Time Frame: Baseline (Day 1) and Week 8
Population: MITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ADS-5102 (260 mg) | ADS-5102 (340 mg) | ADS-5102 (420 mg)
Number analyzed (Participants) | 22 | 19 | 20 | 19
units on a scale | -1.2 (3.08) | 0.0 (3.22) | -3.4 (3.31) | 0.5 (3.23)
Statistical Analysis 1: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.6355, ANCOVA; Least Squares Mean Difference = -2.2, 95% CI 2-sided [-11.2 to 6.9]
Statistical Analysis 2: Comparison: ADS-5102 (420 mg); Test type: Superiority; p = 0.7053, ANCOVA; Least Squares Mean Difference = 1.7, 95% CI 2-sided [-7.2 to 10.6]
Statistical Analysis 3: Comparison: ADS-5102 (260 mg); Test type: Superiority; p = 0.7862, ANCOVA; Change from baseline is a dependent variable, treatment group is a factor, and the baseline value is a covariate; Least Squares Mean Difference = 1.2, 95% CI 2-sided [-7.7 to 10.1]

6. Secondary Outcome: Clinician's Global Impression of Change (CGI-C) in Overall PD Symptoms From Baseline to Week 8
Description: The CGI-C consisted of a single question that assessed the investigator's global impression of the subject's change from Baseline in overall PD symptoms, including but not limited to LID. The CGI-C required that the investigator rate the extent to which the subject's PD had improved or worsened (from marked worsening to marked improvement).
Time Frame: Baseline (Day 1) and Week 8
Population: MITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ADS-5102 (260 mg) | ADS-5102 (340 mg) | ADS-5102 (420 mg)
Number analyzed (Participants) | 22 | 19 | 20 | 19
Participants
  Marked Improvement | 1 | 2 | 7 | 4
  Moderate Improvement | 6 | 8 | 8 | 6
  Minimal Improvement | 4 | 5 | 1 | 5
  No Change | 10 | 3 | 4 | 2
  Minimal Worsening | 1 | 1 | 0 | 0
  Moderate Worsening | 0 | 0 | 0 | 2
  Marked Worsening | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.0036, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: ADS-5102 (420 mg); Test type: Superiority; p = 0.2158, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: ADS-5102 (260 mg); Test type: Superiority; p = 0.1042, Cochran-Mantel-Haenszel; Equally spaced scores

ADVERSE EVENTS:
Time Frame: Baseline through Week 8
Description: The reporting threshold of 5% for Other (Not Including Serious) AEs reflects events that occurred at 5% or greater in any treatment arm.
Arm/Group | Placebo | ADS-5102 (260 mg) | ADS-5102 (340 mg) | ADS-5102 (420 mg)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/20 | 0/21 | 4/20
Other Adverse Events (participants affected / at risk) | 18/22 | 16/20 | 20/21 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | ADS-5102 (260 mg) (N=20) | ADS-5102 (340 mg) (N=21) | ADS-5102 (420 mg) (N=20)
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Mental Status Change (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | ADS-5102 (260 mg) (N=20) | ADS-5102 (340 mg) (N=21) | ADS-5102 (420 mg) (N=20)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 1 | 1
Altered visual depth perception (Eye disorders) | 0 | 0 | 0 | 2
Dry eye (Eye disorders) | 0 | 1 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 7 | 5 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 4 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 2 | 2
Asthenia (General disorders) | 1 | 0 | 3 | 1
Malaise (General disorders) | 0 | 1 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 3 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 2 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 0
Blood glucose increased (Investigations) | 0 | 0 | 2 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 1 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 6 | 3
Headache (Nervous system disorders) | 1 | 1 | 3 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 1 | 1
Somnolence (Nervous system disorders) | 2 | 0 | 1 | 2
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 3 | 3 | 2
Confusional state (Psychiatric disorders) | 1 | 1 | 3 | 2
Hallucination (Psychiatric disorders) | 0 | 1 | 2 | 2
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 2 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 2 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Orthostatic hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No